CLINICAL TRIAL: NCT02066298
Title: Steroids In Eosinophil Negative Asthma
Acronym: SIENA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 007; 1U10HL098115 (NIH)
Record Dates: First submitted 2014-02-10; First posted 2014-02-19 (Estimated); Results first posted 2019-04-18 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: Asthma; Mometasone; Tiotropium
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Mometasone then Tiotropium then Placebo (Experimental): Mometasone 220mcg BID, followed by Tiotropium Respimat 5mcg QD, followed by Placebo
  Interventions: Drug: Mometasone 220mcg BID; Drug: Tiotropium Respimat 5mcg QD; Drug: Placebo
- Mometasone then Placebo then Tiotropium (Experimental): Mometasone 220mcg BID, followed by Placebo, followed by Tiotropium Respimat 5mcg QD
  Interventions: Drug: Mometasone 220mcg BID; Drug: Tiotropium Respimat 5mcg QD; Drug: Placebo
- Placebo then Mometasone then Tiotropium (Experimental): Placebo, followed by Mometasone 220mcg BID, followed by Tiotropium Respimat 5mcg QD
  Interventions: Drug: Mometasone 220mcg BID; Drug: Tiotropium Respimat 5mcg QD; Drug: Placebo
- Placebo then Tiotropium then Mometasone (Experimental): Placebo, followed by Tiotropium Respimat 5mcg QD, followed by Mometasone 220mcg BID
  Interventions: Drug: Mometasone 220mcg BID; Drug: Tiotropium Respimat 5mcg QD; Drug: Placebo
- Tiotropium then Placebo then Mometasone (Experimental): Tiotropium Respimat 5mcg QD, followed by Placebo, followed by Mometasone 220mcg BID
  Interventions: Drug: Mometasone 220mcg BID; Drug: Tiotropium Respimat 5mcg QD; Drug: Placebo
- Tiotropium then Mometasone then Placebo (Experimental): Tiotropium Respimat 5mcg QD, followed by Mometasone 220mcg BID, followed by Placebo
  Interventions: Drug: Mometasone 220mcg BID; Drug: Tiotropium Respimat 5mcg QD; Drug: Placebo

INTERVENTIONS:
Drug: Mometasone 220mcg BID — Mometasone is an ICS
  Other Names: Asmanex
Drug: Tiotropium Respimat 5mcg QD — Tiotropium is a LMA
Drug: Placebo

SUMMARY:
Because approximately half of all mild-moderately-severe asthma is persistently non-eosinophilic, it is important to determine prospectively if patients who are persistently non-eosinophilic differ in their benefit from inhaled corticosteroid treatment compared to patients who are not persistently non-eosinophilic.

DETAILED DESCRIPTION:
SIENA is a 42-week randomized, stratified, 3-period double-blind placebo-controlled crossover study of patients with symptomatic mild-to-moderate asthma, not already taking an inhaled corticosteroid, in whom the effect of "medium-dose" inhaled corticosteroid (ICS) will be compared with the effect of placebo and with a long-acting muscarinic antagonist (LMA).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma for at least previous 12 months.
* Able to perform reproducible spirometry.
* Baseline FEV1≥70% of predicted.
* Asthma confirmed either by:

  * Beta-agonist reversibility to 4 puffs albuterol ≥ 12% OR
  * Methacholine PC20 ≤ 16 mg/ml
* At least 1 of the following indications for chronic controller therapy:

  * Asthma Symptoms > 2 days/week OR
  * Nocturnal Asthma Symptoms > 2 nights/month OR
  * Short-acting beta-agonist use for symptom control > 2 days/week
* For participants ≥18 years of age: Ability to provide informed consent. For participants under 18 years of age: Ability to provide verbal or written assent and ability of parent to provide informed consent.
* Willingness, if female and able to conceive, to utilize one medically-acceptable form of contraception.

Exclusion Criteria:

* Chronic inhaled or oral corticosteroid therapy.
* Use of inhaled or oral corticosteroid therapy within 6 weeks.
* New allergen immunotherapy within the past 3 months or anticipated changes to an ongoing immunotherapy regimen.
* Use of omalizumab within 3 months.
* History of:

  * bladder-neck obstruction, urinary retention or benign prostatic hyperplasia
  * narrow angle glaucoma
  * significant cardiovascular disorders and arrhythmias
  * life-threatening asthma requiring treatment with intubation or mechanical ventilation within the past 5 years
* Respiratory tract infection within past 6 weeks.
* History of smoking within the past 1 year, or > 10 pack-years total if ≥ 18 years of age, or > 5 pack-years total if < 18 years of age.
* Chronic diseases or medical conditions (other than asthma) that could put the participant at risk by participation, e.g. chronic diseases of the lung (other than asthma), heart, liver, kidney, endocrine or nervous system, or immunodeficiency.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, M.D., Study Chair — University of Wisconsin, Madison
Locations (25):
- United States (25):
  - University of Arizona College of Medicine, Tucson, Arizona
  - UCSF Benioff Children's Hospital, San Francisco, California
  - University of California at San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Ann and Robert H. Lurie Children's Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, Case Western Reserve University, Cleveland, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Covar R, Lazarus SC, Krishnan JA, Blake KV, Sorkness CA, Dyer AM, Lang JE, Lugogo NL, Mauger DT, Wechsler ME, Wenzel SE, Cardet JC, Castro M, Israel E, Phipatanakul W, King TS; National Heart, Lung, and Blood Institute AsthmaNet. Association of Sputum Eosinophilia With Easily Measured Type-2 Inflammatory Biomarkers in Untreated Mild Persistent Asthma. J Allergy Clin Immunol Pract. 2024 Apr;12(4):960-969.e6. doi: 10.1016/j.jaip.2023.12.010. Epub 2023 Dec 12. PMID 38097180
- [Derived] Lazarus SC, Krishnan JA, King TS, Lang JE, Blake KV, Covar R, Lugogo N, Wenzel S, Chinchilli VM, Mauger DT, Dyer AM, Boushey HA, Fahy JV, Woodruff PG, Bacharier LB, Cabana MD, Cardet JC, Castro M, Chmiel J, Denlinger L, DiMango E, Fitzpatrick AM, Gentile D, Hastie A, Holguin F, Israel E, Jackson D, Kraft M, LaForce C, Lemanske RF Jr, Martinez FD, Moore W, Morgan WJ, Moy JN, Myers R, Peters SP, Phipatanakul W, Pongracic JA, Que L, Ross K, Smith L, Szefler SJ, Wechsler ME, Sorkness CA; National Heart, Lung, and Blood Institute AsthmaNet. Mometasone or Tiotropium in Mild Asthma with a Low Sputum Eosinophil Level. N Engl J Med. 2019 May 23;380(21):2009-2019. doi: 10.1056/NEJMoa1814917. Epub 2019 May 19. PMID 31112384
- [Derived] Sorkness CA, King TS, Dyer AM, Chinchilli VM, Mauger DT, Krishnan JA, Blake K, Castro M, Covar R, Israel E, Kraft M, Lang JE, Lugogo N, Peters SP, Wechsler ME, Wenzel SE, Lazarus SC; National Heart Lung and Blood Institute's "AsthmaNet". Adapting clinical trial design to maintain meaningful outcomes during a multicenter asthma trial in the precision medicine era. Contemp Clin Trials. 2019 Feb;77:98-103. doi: 10.1016/j.cct.2018.12.012. Epub 2018 Dec 27. PMID 30593883
- See also: AsthmaNet — http://asthmanetresearch.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Then Tiotropium Then Placebo: Mometasone 220mcg BID, followed by Tiotropium Respimat 5mcg QD, followed by Placebo
  Mometasone 220mcg BID: Mometasone is an ICS
  Tiotropium Respimat 5mcg QD: Tiotropium is a LMA
  Placebo
- Mometasone Then Placebo Then Tiotropium: Mometasone 220mcg BID, followed by Placebo, followed by Tiotropium Respimat 5mcg QD
  Mometasone 220mcg BID: Mometasone is an ICS
  Tiotropium Respimat 5mcg QD: Tiotropium is a LMA
  Placebo
- Placebo Then Mometasone Then Tiotropium: Placebo, followed by Mometasone 220mcg BID, followed by Tiotropium Respimat 5mcg QD
  Mometasone 220mcg BID: Mometasone is an ICS
  Tiotropium Respimat 5mcg QD: Tiotropium is a LMA
  Placebo
- Placebo Then Tiotropium Then Mometasone: Placebo, followed by Tiotropium Respimat 5mcg QD, followed by Mometasone 220mcg BID
  Mometasone 220mcg BID: Mometasone is an ICS
  Tiotropium Respimat 5mcg QD: Tiotropium is a LMA
  Placebo
- Tiotropium Then Placebo Then Mometasone: Tiotropium Respimat 5mcg QD, followed by Placebo, followed by Mometasone 220mcg BID
  Mometasone 220mcg BID: Mometasone is an ICS
  Tiotropium Respimat 5mcg QD: Tiotropium is a LMA
  Placebo
- Tiotropium Then Mometasone Then Placebo: Tiotropium Respimat 5mcg QD, followed by Mometasone 220mcg BID, followed by Placebo
  Mometasone 220mcg BID: Mometasone is an ICS
  Tiotropium Respimat 5mcg QD: Tiotropium is a LMA
  Placebo
Period: Overall Study
Arm/Group | Mometasone Then Tiotropium Then Placebo | Mometasone Then Placebo Then Tiotropium | Placebo Then Mometasone Then Tiotropium | Placebo Then Tiotropium Then Mometasone | Tiotropium Then Placebo Then Mometasone | Tiotropium Then Mometasone Then Placebo
Started | 49 | 48 | 50 | 51 | 47 | 50
Completed 1st Period | 44 | 47 | 45 | 48 | 46 | 45
Completed 2nd Period | 41 | 41 | 41 | 46 | 42 | 41
Completed 3rd Period | 40 | 40 | 40 | 45 | 38 | 38
Completed | 40 | 40 | 40 | 45 | 38 | 38
Not Completed | 9 | 8 | 10 | 6 | 9 | 12
Not completed — Lost to Follow-up | 3 | 2 | 3 | 2 | 3 | 4
Not completed — Withdrawal by Subject | 6 | 6 | 6 | 4 | 5 | 8
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Then Tiotropium Then Placebo | Mometasone Then Placebo Then Tiotropium | Placebo Then Mometasone Then Tiotropium | Placebo Then Tiotropium Then Mometasone | Tiotropium Then Placebo Then Mometasone | Tiotropium Then Mometasone Then Placebo | Total
Number analyzed (Participants) | 49 | 48 | 50 | 51 | 47 | 50 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (15.3) | 32.6 (13.8) | 33.2 (13.9) | 30.0 (14.8) | 30.8 (12.5) | 28.2 (12.9) | 31.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 32 | 33 | 27 | 33 | 184
  Male | 20 | 18 | 18 | 18 | 20 | 17 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 4 | 7 | 7 | 7 | 35
  Not Hispanic or Latino | 43 | 44 | 46 | 44 | 40 | 43 | 260
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 3 | 0 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 14 | 15 | 16 | 14 | 16 | 88
  White | 34 | 32 | 33 | 31 | 32 | 30 | 192
  More than one race | 0 | 0 | 0 | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 48 | 50 | 51 | 47 | 50 | 295
Forced expiratory volume at one second (FEV1) Percent of Predicted [Mean (Standard Deviation); unit: percentage of predicted FEV1] — FEV1, expressed as percent of predicted FEV1 based on age, sex, race, and height.
  percentage of predicted FEV1 | 90.6 (11.5) | 91.5 (11.2) | 92.0 (11.8) | 93.8 (12.4) | 91.7 (13.6) | 91.6 (12.5) | 91.9 (12.1)
Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Asthma Control Test: The score is calculated as the sum total of a 5-item questionnaire. Each item ranges from 1 (poor control) to 5 (good control) so that the range of the total score is 5 to 25. Scores below 20 indicate that asthma is not well controlled.
  units on a scale | 21.3 (2.3) | 21.2 (2.5) | 21.1 (2.7) | 20.9 (2.2) | 20.9 (2.8) | 21.1 (2.5) | 21.1 (2.5)
Sputum differential count - Percent eosinophils [Median (Inter-Quartile Range); unit: percentage of cells] — Percentage of cells collected from induced sputum that are eosinophils
  percentage of cells | 0.1 [0.0 to 0.4] | 0.4 [0.0 to 1.7] | 0.4 [0.0 to 2.4] | 0.2 [0.0 to 1.0] | 0.2 [0.0 to 0.7] | 0.2 [0.0 to 0.8] | 0.2 [0.0 to 1.0]
Blood differential count - Percent eosinophils [Median (Inter-Quartile Range); unit: percentage of cells] — Percentage of blood cells that are eosinophils
  percentage of cells | 2.3 [1.1 to 4.1] | 4.0 [2.0 to 5.3] | 3.0 [1.9 to 4.7] | 3.2 [2.0 to 5.0] | 3.0 [1.5 to 5.0] | 2.8 [1.0 to 4.0] | 3.0 [1.7 to 5.0]

OUTCOME MEASURES:

1. Primary Outcome: Pairwise Comparison of Treatments Based on Composite Measure Using Treatment Failures, Asthma Control Days, and Percent Predicted FEV1.
Description: This composite outcome uses a hierarchical method to ascertain differences in asthma control. For each participant, treatments are first compared to see if they differ in terms of treatment failures. If one treatment results in no treatment failures and another treatment does, it is deemed the superior treatment and no further comparisons are made. If treatment superiority cannot be assigned by treatment failures, then they are compared by asthma control days (ACDs). If one treatment yields at least 31 annualized ACDs more than another, it is deemed the superior treatment. If treatment superiority still cannot be assigned by ACDs, then they are compared by percent predicted FEV1 at the end of a treatment period. If one treatment yields at least 5% greater FEV1 than another, it is deemed the superior treatment. If treatment superiority cannot be assigned by exacerbations, ACDs or FEV1, then that participant is classified as having no differential response.
Time Frame: End of 12-week treatment period
Population: For each pairwise comparison (mometasone vs. placebo and tiotropium vs. placebo), participants were required to complete both of the relevant treatment periods in order to be included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Eosinophil Low: Participants with sputum eosinophils < 2% at study entry
- Eosinophil High: Participants with sputum eosinophils >= 2% at study entry
Arm/Group | Eosinophil Low | Eosinophil High
Number analyzed (Participants) | 184 | 67
Participants
  Mometesone superior to placebo: number analyzed (Participants) | 176 | 67
  Mometesone superior to placebo | 74 | 35
  Placebo superior to mometasone: number analyzed (Participants) | 176 | 67
  Placebo superior to mometasone | 56 | 12
  Mometesone equal to placebo: number analyzed (Participants) | 176 | 67
  Mometesone equal to placebo | 46 | 20
  Tiotropium superior to placebo: number analyzed (Participants) | 181 | 62
  Tiotropium superior to placebo | 80 | 25
  Placebo superior to tiotropium: number analyzed (Participants) | 181 | 62
  Placebo superior to tiotropium | 52 | 19
  Tiotropium equal to placebo: number analyzed (Participants) | 181 | 62
  Tiotropium equal to placebo | 49 | 18
Statistical Analysis 1: Comparison: Eosinophil Low; The null hypothesis was that, among those participants for which either mometasone is not equal to placebo, the proportion for which mometasone is superior to placebo is equal to the proportion for which placebo is superior to mometasone. The trial was designed to provide power of 0.85 for a 0.20 difference between the proportions being compared at a significance level of 0.025; Test type: Superiority; p = 0.14, exact binomial test; a priori threshold for significance was 0.025
Statistical Analysis 2: Comparison: Eosinophil Low; The null hypothesis was that, among those participants for which either tiotropium is not equal to placebo, the proportion for which tiotropium is superior to placebo is equal to the proportion for which placebo is superior to tiotropium. The trial was designed to provide power of 0.85 for a 0.20 difference between the proportions being compared at a significance level of 0.025; Test type: Superiority; p = 0.029, exact binomial test — a priori threshold for significance was 0.025
Statistical Analysis 3: Comparison: Eosinophil High; The null hypothesis was that, among those participants for which either mometasone is not equal to placebo, the proportion for which mometasone is superior to placebo is equal to the proportion for which placebo is superior to mometasone. This was an exploratory analysis and there were no power considerations; Test type: Superiority; p = 0.001, exact binomial test — this analysis is considered exploratory
Statistical Analysis 4: Comparison: Eosinophil High; The null hypothesis was that, among those participants for which either tiotropium is not equal to placebo, the proportion for which tiotropium is superior to placebo is equal to the proportion for which placebo is superior to tiotropium. This was an exploratory analysis and there were no power considerations; Test type: Superiority; p = 0.45, exact binomial test — this analysis is considered exploratory

2. Secondary Outcome: Treatment Failure
Description: Treatment Failure includes:
  * Awakening from asthma three or more times in a two-week period or on two consecutive nights, or
  * Using albuterol for relief of symptoms four or more times/day for two or more consecutive days, or
  * Albuterol has been relieving symptoms for less than four hours after each treatment over a 12-hour period, or
  * Using albuterol for relief of symptoms daily for seven days, and this use exceeds two times the weekly use of albuterol in the baseline period, or
  * exercise induces unusual breathlessness
Time Frame: End of 12-week treatment period
Population: participants who completed the treatment period with data to evaluate treatment failure outcome
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: The placebo treatment period for all participants.
- Mometasone 220mcg BID: The mometasone treatment period for all participants. Mometasone administered 220mcg BID
- Tiotropium Respimat 5mcg QD: The tiotropium treatment period for all participants. Tiotropium administered 5mcg QD
Arm/Group | Placebo | Mometasone 220mcg BID | Tiotropium Respimat 5mcg QD
Number analyzed (Participants) | 254 | 255 | 258
Participants | 29 | 29 | 35

3. Secondary Outcome: Annualized Asthma Control Days
Description: Asthma Control Days (ACD) are based on patient completed electronic daily diaries, and are defined as: A day with no rescue albuterol use (pre-exercise albuterol will not be counted), no non-study asthma medications, no daytime asthma symptoms (shortness of breath, wheezing, chest tightness, phlegm/mucus rated as mild, moderate or severe, or cough rated as moderate or severe), no nighttime asthma symptoms, no unscheduled healthcare visits for asthma, and no PEF < 80% of predetermined baseline. Annualized ACD are calculated as the proportion of ACD during the treatment period multiplied by 365.
Time Frame: End of 12-week treatment period
Population: participants who completed the treatment period with data to evaluate asthma control days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Mometasone 220mcg BID | Tiotropium Respimat 5mcg QD
Number analyzed (Participants) | 216 | 225 | 228
days | 179 (137) | 186 (141) | 176 (139)

4. Secondary Outcome: Forced Expiratory Volume at One Second (FEV1) Percent of Predicted
Description: FEV1, expressed as percent of predicted FEV1 based on age, sex, race, and height.
Time Frame: End of 12-week treatment period
Population: participants who completed the treatment period and were able to provide FEV1 measurements
Measure: Mean (Standard Deviation); unit: percentage of predicted FEV1
Groups:
- Eosinophil Low - Placebo: The placebo treatment period for all participants
Arm/Group | Eosinophil Low - Placebo | Mometasone 220mcg BID | Tiotropium Respimat 5mcg QD
Number analyzed (Participants) | 254 | 247 | 252
percentage of predicted FEV1 | 92 (14) | 94 (13) | 95 (14)

5. Secondary Outcome: Peak Expiratory Flow Rate
Description: Peak expiratory flow rate is a person's maximum speed of expiration. It measures the airflow through the bronchi and thus the degree of obstruction in the airways.
Time Frame: End of 12-week treatment period
Population: participants who completed the treatment period and were able to provide FEV1 measurements
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Placebo | Mometasone 220mcg BID | Tiotropium Respimat 5mcg QD
Number analyzed (Participants) | 253 | 249 | 256
liters per minute | 476 (117) | 485 (117) | 497 (117)

6. Secondary Outcome: Asthma Exacerbations
Description: Asthma exacerbations are more severe episodes of acute worsening, defined by meeting one or more of the following:
  * FEV1 <50% of baseline on 2 consecutive measurements
  * FEV1 <40% of predicted on 2 consecutive measurements
  * Use of ≥ 16 puffs of "as needed" β-agonist per 24 hours for a period of 48 hours
  * Use of oral/parenteral corticosteroid due to asthma
Time Frame: End of 12-week treatment period
Population: participants who completed the treatment period with data to evaluate exacerbations
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Mometasone 220mcg BID | Tiotropium Respimat 5mcg QD
Number analyzed (Participants) | 254 | 255 | 258
Participants | 1 | 3 | 5

ADVERSE EVENTS:
Time Frame: Each participant was followed over the course of three 12-week treatment periods for a total of 36 weeks. The adverse events recorded below are reported at the treatment period level and represent 12 weeks of "at risk" exposure time.
Arm/Group | Placebo | Mometasone 220mcg BID | Tiotropium Respimat 5mcg QD
All-Cause Mortality (participants affected / at risk) | 0/276 | 0/275 | 0/271
Serious Adverse Events (participants affected / at risk) | 0/276 | 6/275 | 2/271
Other Adverse Events (participants affected / at risk) | 45/276 | 47/275 | 38/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=276) | Mometasone 220mcg BID (N=275) | Tiotropium Respimat 5mcg QD (N=271)
pregnancy (Pregnancy, puerperium and perinatal conditions) | NA | 1 (1) | 0 (0)
closed fracture of lower end of humerus (Musculoskeletal and connective tissue disorders) | NA | 1 (1) | 0 (0)
Partial bowel obstruction. (Gastrointestinal disorders) | NA | 0 (0) | 1 (1)
Hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 (0) | 1 (1)
Unspecified nonpsychotic mental disorder (Psychiatric disorders) | NA | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | NA | 1 (1) | 0 (0)
malignant neoplasm of skin of other and unspecified parts of face (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 (1) | 0 (0)
Acute appendicitis without mention of peritonitis (Gastrointestinal disorders) | NA | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=276) | Mometasone 220mcg BID (N=275) | Tiotropium Respimat 5mcg QD (N=271)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 37 (42) | 33 (38) | 29 (37)
Acute URI not otherwise specified (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 16 (18) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT02066298/Prot_SAP_000.pdf